CLINICAL TRIAL: NCT01065441
Title: A Phase I/II Study of an Experimental Therapeutic Cancer Vaccine Created In-situ in Patients With Stage II-Stage IV Cancers
Brief Title: Experimental Therapeutic Cancer Vaccine Created In-situ in Patients With Stage II-Stage IV Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael Har-Noy (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor-Investigator, Michael Har-Noy, Investigator: Dept of Bone Marrow Transplantation and Immunotherapy, Mirror Biologics, Inc.
Organization: Mirror Biologics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-002-HMC
Record Dates: First submitted 2010-02-07; First posted 2010-02-09 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumors Stage II, Stage III and Stage IV; Breast Cancer; Colorectal Cancer; Prostate Cancer; Melanoma; Ovarian Cancer; Sarcoma; Non-small Cell Lung Cancer
Keywords: breast cancer; colorectal cancer; prostate cancer; melanoma; ovarian cancer; GI cancer; Sarcoma; Renal Cell Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Melanoma; Ovarian Neoplasms; Sarcoma; Carcinoma, Non-Small-Cell Lung; Gastrointestinal Neoplasms; Carcinoma, Renal Cell | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: AlloStim — Patients meeting eligibility criteria will be primed with at least three and up to nine intradermal AlloStim-TM injections at a frequency of every 2-8 days at doses between 1-4 x 10^7 cells
Procedure: Cryoablation — Percutaneous cryoablation of selected tumor lesion under CT or US guidance
Biological: AlloStim — intratumoral injection of AlloStim-TM into cryoablated tumor lesion at a dose of 1-6 x 10^7 cells
Biological: AlloStim — intravenous AlloStim-TM at doses between 1 x 10^7 to 1 x 10^9 cells
Biological: AlloStim — Intraperitoneal AlloStim-TM infusion in patients with peritoneal carcinomatosis and/or ascites
Biological: AlloStim — Patients with malignant pleural effusion may receive intrapleural AlloStim-TM infusion at a dose of 5-10 x 10^7 cells.
Biological: AlloStim — Patients with palpable tumors may receive alcohol ablation and intratumoral AlloStim-TM

SUMMARY:
A Phase I/II study of an in-situ therapeutic cancer vaccine. Vaccines contain a source of antigen and and adjuvant. In this study the source of tumor antigen comes from the killing of a selected tumor by cryoablation (killing using extreme cold) and the adjuvant is intentionally mis-matched immune cells (AlloStim-TM) engineered to produce inflammatory cytokines.

DETAILED DESCRIPTION:
This is a Phase I/II clinical study to investigate the optimal protocol and indication for creating a personalized anti-tumor vaccine within the body of patients with cancer. The aim of the study is to evaluate the safety of administration and anti-tumor effect of a vaccine protocol that has three separate steps. Cancer patients generally present with an immune response to cancer biased to a Th2 response, while a Th1 response is considered necessary for mediating anti-tumor immunity. The first step of the study consists of multiple intradermal priming doses of AlloStimTM. The aim of this step is to create Th1 immunity to the alloantigens in AlloStimTM, thus increasing the number of Th1 cells in circulation. The second step of the protocol involves the cryoablation of a selected tumor lesion followed by an intratumoral AlloStimTM injection. The aim of this step is to generate tumor-specific CTL killer cells in the circulation. The final step is an intravenous infusion of AlloStimTM. The aim of this step is to activate circulating Th1 cells, killer cells, and natural killer cells. The further aim of this step is to create an inflammatory environment that can break-down the ability of the tumor to avoid an anti-tumor immune response. In patients with partial responses and recurrence of disease, additional intravenous "booster" infusions are utilized to reactivate the circulating immune cells.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Stage II-IV including breast cancer, colorectal cancer, non-small cell lung cancer, ovarian or other gynecological cancer, prostate cancer, pancreatic or other GI cancer, melanoma, head or neck cancer or lymphoma/plasmacytoma.
* Measurable disease determined upon review of abdominal and/or chest CT scan within 60 days of evaluation for study inclusion with a target tumor lesion for cryoablation or alcohol ablation located in liver, kidney, bone, lung, adrenal, pancreas, lymph node, skin, neck or prostate deemed to be accessible for percutaneous access or carcinomatosis or malignant ascites or malignant pleural effusion.
* When applicable, acceptable cryoablation procedure technique risk: the target tumor for ablation must have adequate distance from adjacent vasculature and other organs to permit safe application of cryoprobe (generally, more than a 2.5cm clearance of the cryoprobe from any vital structure such as the bowel, inferior vena cava, or aorta). The safety assessment of the cryoprobe placement will be made an attending radiologist based on imaging studies.
* Life expectancy >90 days
* No bevacizumab (Avastin®) within 6 weeks of planned cryoablation procedure
* ECOG status 0-2
* No concurrent medication known to interfere with platelet function or coagulation (e.g., aspirin, ibuprofen, clopidogrel, or warfarin) unless such medications can be discontinued for an appropriate time period based on the drug half-life and known activity (e.g., aspirin for 7 days) prior to cryoablation procedure
* No low molecular weight heparin preparations unless can be discontinued 8 hours prior to cryoablation
* At least 2 weeks since prior cytotoxic chemotherapy
* Absolute granulocyte count ≥ 1,200/mm3
* Platelet count ≥ 100,000/mm3
* PT/INR ≤ 1.5

  o INR correctable to ≤ 1.5 or a PT/PTT correctable to normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be monitored weekly prior to the cryoablation day to assure INR is stable. However, heparin or warfarin must be withheld prior to cryoablation such that the above criteria are met.
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 times normal
* Alkaline phosphatase ≤ 2.5 times normal (≤ 5 times normal if liver involvement)
* Aspartate aminotransferase (AST) or (SGOT) ≤ 2.5 times ULN
* Alanine aminotransferase (ALT) or (SGPT) ≤ 2.5 times ULN
* Not pregnant or lactating
* Patients with child bearing potential must agree to use adequate contraception
* No psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation
* Study specific informed consent

Exclusion Criteria:

* Taking anticoagulant medication for concomitant medical condition (unless can be safely discontinued for cryoablation procedure)
* Prior allogeneic bone marrow/stem cell or solid organ transplant
* Chronic use (> 2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to > 10 mg/day of prednisone) within 30 days of the first day of study drug treatment

  o Topical and inhaled corticosteroids are permitted
* Concomitant active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis)
* Prior experimental cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine)
* Immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 3 months of study entry
* History of blood transfusion reactions
* Known allergy to bovine products
* Know allergy to murine products
* Progressive viral or bacterial infection

  o All infections must be resolved and the patient must remain afebrile for seven days without antibiotics prior to being placed on study
* Cardiac disease of symptomatic nature or cardiac ejection fraction < 45%
* Symptomatic pulmonary disease or FEV1, FVC, and DLCO ≤ 50% predicted
* History of HIV positivity or AIDS o HBV and/or HCV positivity is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the evaluation of any drug-related toxicity associated with AlloStimTM administration as well as the reversibility of such toxicity. | 90 days

SECONDARY OUTCOMES:
The secondary end-point is the evaluation of the anti-tumor effect of AlloStimTM administration. | 1 year
The tertiary end-point is the evaluation of the immunological response to AlloStim-TM administration. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Peretz, MD, Principal Investigator — Hadassah Medical Organization; Dr. Michael Har-Noy, Study Chair — Mirror Biologics, Inc.
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Background] Har-Noy M, Zeira M, Weiss L, Slavin S. Completely mismatched allogeneic CD3/CD28 cross-linked Th1 memory cells elicit anti-leukemia effects in unconditioned hosts without GVHD toxicity. Leuk Res. 2008 Dec;32(12):1903-13. doi: 10.1016/j.leukres.2008.05.007. Epub 2008 Jun 18. PMID 18565579
- [Background] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441